CLINICAL TRIAL: NCT01910987
Title: A Randomized, Controlled Phase 3 Study to Evaluate Optimized Retreatment and Prolonged Therapy With Bortezomib (Velcade) in Patients With Multiple Myeloma in First or Second Relapse.
Brief Title: Study to Evaluate Optimized Retreatment and Prolonged Therapy With Bortezomib
Acronym: OPTIMRETREAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR018796; 26866138MMY3033 (Other: Janssen-Cilag International NV); 2011-004795-11 (EudraCT Number)
Record Dates: First submitted 2013-02-04; First posted 2013-07-30 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; bortezomib; Velcade; First or Second Relapse; retreatment; Prolonged therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- optimized retreatment, prolonged therapy (Experimental): Patients will start therapy with retreatment with 6 cycles of bortezomib and dexamethasone (two 21-day cycles followed by four 35-day cycles) followed by a second randomization in a 1:1 ratio to 1 of 2 prolonged therapy schedules with bortezomib alone (Group A1: once weekly for the first 4 weeks in 35-day cycles; or Group A2: once every other week)
  Interventions: Drug: bortezomib (optimized retreatment); Drug: dexamethasone (optimized retreatment)
- standard retreatment (Other): Current Standard of Care: Patients will start retreatment with eight 21-day bortezomib and dexamethasone cycles, followed by posttreatment follow-up every 6 weeks.
  Interventions: Drug: bortezomib (standard retreatment); Drug: dexamethasone (standard retreatment)

INTERVENTIONS:
Drug: bortezomib (optimized retreatment) — Type= exact number, unit = mg/m2 body surface area, number = 1.3, form = powder for solution for injection, route = subcutaneous, injection on Days 1, 4, 8 and 11, every 21 days of cycle 1 and 2; injection on Days 1, 8, 15, 22, every 35 days for cycles 3 to 6; followed by injections on Days 1, 8, 15, 22 every 35 days (Group A1) or injections every other week (Group A2). Treatment will be stopped at confirmed disease progression
  Arms: optimized retreatment, prolonged therapy
Drug: dexamethasone (optimized retreatment) — Type= exact number, unit = mg, number = 20, form = tablet, route = oral, intake on Days 1, 2, 4, 5, 8, 9, 11 and 12, every 21 days of cycle 1 and 2; intake on Days 1, 2, 8, 9, 15, 16, 22 and 23 every 35 days for cycles 3 to 6
  Arms: optimized retreatment, prolonged therapy
Drug: bortezomib (standard retreatment) — Type= exact number, unit = mg/m2 body surface area, number = 1.3, form = powder for solution for injection, route = subcutaneous, injection on Days 1,4,8,11, every 21 days for cycles 1 to 8 or until confirmed disease progression
  Arms: standard retreatment
Drug: dexamethasone (standard retreatment) — Type = exact number, unit = mg, number = 20, form = tablet, route= oral, intake on Days 1, 2, 4, 5, 8, 9, 11, 12, every 21 days for cycles 1 to 8 or until confirmed disease progression
  Arms: standard retreatment

SUMMARY:
The objective of this study is to describe the effect of optimized retreatment with bortezomib in combination with dexamethasone followed by prolonged therapy with bortezomib, versus standard retreatment with bortezomib in combination with dexamethasone on progression free survival (PFS).

DETAILED DESCRIPTION:
This is an interventional, randomized (assignment to a group is happening by chance, like flipping a coin), open-label, parallel-group, event-driven, international, multicenter, Phase 3 study. This study has different phases: a pre-treatment phase, a treatment phase (which consists of an optimized retreatment period followed by a prolonged therapy period, or a standard retreatment period followed by a posttreatment period), and a long-term follow-up phase for survival up to the end of the study. Before the premature stopping of enrollment, the end of the study was event-driven, defined as 1 year after 186 events (an 'event' being defined as disease progression or death). Following the premature stopping of enrollment, effective 20 June 2014, the end of the study is defined as a maximum of 18 months after enrollment of the last patient in the study. After providing written informed consent, patients will be evaluated for eligibility during a 14-day pre-treatment period. The study doctor will carry out tests to see if the patient is suitable for this study, within the two weeks before receipt of the first dose of the study drugs. Once it has been determined that the patient is able to participate, he/she will be randomly assigned to 1 of 2 different bortezomib retreatment schedules. In this first randomization, patients will receive optimized retreatment or standard retreatment in a 2:1 ratio. Group A: optimized retreatment followed by prolonged therapy. Patients will start therapy with retreatment with 6 cycles of bortezomib and dexamethasone (two 21-day cycles followed by four 35-day cycles) followed by a second randomization in a 1:1 ratio to 1 of 2 prolonged therapy schedules with bortezomib alone (Group A1: once weekly for the first 4 weeks in 35-day cycles; or Group A2: once every other week). Group B: standard retreatment with eight 21-day bortezomib and dexamethasone cycles, followed by posttreatment follow-up every 6 weeks. During the retreatment phase, a series of tests will be done at the first day of each cycle. For patients in Group A the doctor will assess if the patient has responded to the treatment or not. Only if the patient responded, will he/she be able to continue in the prolonged therapy part of the study. At this time the patient will be randomized to one of the two groups (Group A1 or Group A2) in the prolonged therapy phase. During the prolonged therapy phase the disease status and the response to therapy will be evaluated every 6 weeks. This phase will continue until the disease progresses, in case there are unacceptable toxicities despite dose modifications. During the posttreatment period patients in group B will continue to be evaluated for disease status every 6 weeks until confirmed disease progression, when they start alternative multiple myeloma treatment, are withdrawn from the study, death or at the end of the study (a maximum of 18 months after the last patient is enrolled in the study), whichever occurs first. In case the patient discontinues bortezomib before disease progression during the treatment phase, he/she will be asked to complete the End of Study Visit procedures and will be evaluated every 6 weeks until confirmed disease progression, when they start alternative multiple myeloma treatment, are withdrawn from the study, death or at the end of the study (a maximum of 18 months after the last patient is enrolled in the study), whichever occurs first. All patients will have an End of Trial Visit performed 30 to 35 days after the last administration of bortezomib, or as soon as possible after bortezomib treatment is discontinued for patients receiving alternative multiple myeloma therapy. After confirmed disease progression or start of the first alternative multiple myeloma therapy, patients will enter the long-term follow-up phase for up to a maximum of 18 months after the last patient is enrolled in the study. During this phase, the patients will be contacted by at least a telephone call every other month to be followed up for the first alternative multiple myeloma therapy and survival. From the end of the study in countries where bortezomib is not commercially available for prolonged therapy or is not accessible (via a national program or access program) at that time, patients who in the opinion of the investigator would continue to benefit from prolonged therapy with bortezomib, will continue to be supplied with bortezomib until it is accessible in that particular country or for a period of 2 years, whichever occurs first. Before the premature stopping of enrollment, it was planned to enroll a target of 240 patients in this study.

ELIGIBILITY:
Inclusion Criteria:

* Have received a bortezomib containing regimen in one of the previous line(s) of therapy and have shown at least PR to the previous bortezomib therapy.
* Have relapsed / progressed multiple myeloma following 1 or 2 previous lines of therapy as defined in the protocol.
* Have measurable secretory multiple myeloma: measurable disease for secretory multiple myeloma is defined by at least one of the following measurements: serum M protein greater than or equal to 1 g/dL (≥10g/L], urine M-protein of ≥200 mg/24 hours.
* Have an ECOG performance status of ≤2.
* Have a life expectancy estimated at screening of ≥6 months.

Exclusion Criteria:

* Has received more than 2 previous lines of therapy for multiple myeloma or has received no previous bortezomib-containing regimen.
* Has been refractory to bortezomib, defined as either having progressed during bortezomib therapy or relapsed/progressed within 6 months after the last dose of bortezomib.
* Has oligosecretory or nonsecretory multiple myeloma.
* Has a history of a myocardial infarction within 6 months of enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Has peripheral neuropathy or neuropathic pain of grade 2 or greater intensity, as defined by the National Cancer Institute Common Terminology Criteria of Adverse Events (NCI CTCAE), version 4.0.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Effect of optimized retreatment followed by prolonged therapy versus standard retreatment on Progression Free Survival (PFS) | follow up to disease progression or death or to a maximum of 18 months after the last patient is enrolled in the study, whichever occurs first
  Time from randomization to therapy to time of diagnosis of PD or death due to any cause

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | at end of treatment (defined as a maximum of 6 months in group B and an expected average of 17 months in group A)
  Overall response rate as defined by the combination of patients with complete response, very good partial response and partial response according to the International Myeloma Working Group 2011 criteria (IMWG)
Time to Progression (TTP) | at end of treatment (defined as a maximum of 6 months in group B and an expected average of 17 months in group A)
  Time to Progression is defined as the time from baseline to PD, discontinuation/withdrawal or death.
Duration of Response (DOR) | at end of treatment (defined as a maximum of 6 months in group B and an expected average of 17 months in group A)
  DOR is defined as the duration from the date of the best confirmed response for patients who achieved Complete Response (CR) or Partial Response (PR) to the date of first documented evidence of PD over the duration of the study.
Time to Next Myeloma Therapy (TTNT) | at end of treatment (defined as a maximum of 6 months in group B and an expected average of 17 months in group A)
Overall Survival (OS) | at end of treatment (defined as a maximum of 6 months in group B and an expected average of 17 months in group A)
Eastern Cooperative Oncology Group (ECOG) Performance Status | at end of treatment (defined as a maximum of 6 months in group B and an expected average of 17 months in group A)
  The ECOG Performance Status is used to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis. The score ranges from 0 "fully active, able to carry on all pre-disease performance without restriction" to 5 "dead".
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - C30 (EORTC QLQ-C30) | at end of treatment (defined as a maximum of 6 months in group B and an expected average of 17 months in group A)
  The EORTC QLQ-C30 incorporates 5 functional scales (physical, role, emotional, cognitive and social functioning), 1 global health and quality of life scale, 3 symptom scales (fatigue, nausea/vomiting and pain), and 6 single items (dyspnoea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The recall period is 1 week (the past week). It is a 30-item questionnaire with responses ranging for the functional scales from not at all to very much and the global health/QOL ranging from very poor to excellent. Scores are transformed to 0-100 scale.
European Quality of Life-5 Dimensions Questionnaire (EQ-5D) | at end of treatment (defined as a maximum of 6 months in group B and an expected average of 17 months in group A)
  The EQ-5D is a 5-item questionnaire and a "thermometer" visual analogue scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state)

CONTACTS AND LOCATIONS:
Locations (54):
- Belgium (7):
  - Antwerp
  - Edegem
  - Haine-Saint-Paul
  - Hasselt
  - Sint-Niklaas
  - Turnhout
  - Yvoir
- Finland (3):
  - Helsinki
  - Lahti
  - Turku
- France (5):
  - Lille
  - Paris
  - Périgueux
  - Rennes
  - Tours
- Germany (6):
  - Cologne
  - Dresden
  - Heidelberg
  - Mutlangen
  - Osnabrück
  - Rostock
- Israel (3):
  - Haifa
  - Nahariya
  - Ramat Gan
- Netherlands (5):
  - Apeldoorn
  - Deventer
  - Heerlen
  - Tilburg
  - Zwolle
- Norway (3):
  - Fredrikstad
  - Stavanger
  - Trondheim
- Poland (8):
  - Brzozów
  - Chorzów
  - Lodz
  - Lublin
  - Olsztyn
  - Opole
  - Słupsk
  - Wroclaw
- Portugal (3):
  - Coimbra
  - Ponta Delgada
  - Porto
- Sweden (4):
  - Borås
  - Falun
  - Huddinge
  - Stockholm
- Turkey (Türkiye) (7):
  - Adana
  - Ankara
  - Bursa
  - Istanbul
  - Izmir
  - Samsun
  - Trabzon

REFERENCES:
- [Derived] Terpos E, Gobbi M, Potamianou A, Lahaye M, Couturier C, Cavo M. Retreatment and prolonged therapy with subcutaneous bortezomib in patients with relapsed multiple myeloma: A randomized, controlled, phase III study. Eur J Haematol. 2018 Jan;100(1):10-19. doi: 10.1111/ejh.12937. Epub 2017 Oct 30. PMID 28801967
- See also: A Randomized, Controlled, Phase 3 Study to Evaluate Optimized Retreatment and Prolonged Therapy With Bortezomib (VELCADE) in Patients With Multiple Myeloma in First or Second Relapse — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=3334&filename=CR018796_EudraCT%20Full%20Data%20Set.pdf